CLINICAL TRIAL: NCT01622894
Title: Genetics of Mendelian Forms of Young Onset Alzheimer Disease. Identification of Novel Genetic Causes of AD Are of Importance in Completing the Mechanisms of the Amyloid Hypothesis. This Project is Useful to Promote the Guidelines on the Genetic Diagnosis of AD in France.
Brief Title: Genetics of Mendelian Forms of Young Onset Alzheimer Disease
Acronym: GMAJ
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2008/067/HP; 2009-010884-18
Record Dates: First submitted 2012-06-14; First posted 2012-06-19 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Autosomal Dominant Cases of Alzheimer 's Disease
Keywords: Alzheimer genetics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — samples with DNA
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Genetics of mendelian forms of young onset Alzheimer Disease (GMAJ project)

Introduction : Autosomal dominant forms of Alzheimer disease (AD) are characterized by young age of onset. In France the prevalence was estimated at around 1000 cases. The Phenotypical Expression: There is diversity in phenotypical expression, associating dementia, spastic paraplegia, early extrapyramidal syndrome, ataxia or stroke caused by severe cerebral amyloid angiopathy. Diversity in neuropathological expression is demonstrated by the presence of cotton wool plaques, Lewy bodies with Lewy neurites and severe cerebral amyloid angiopathy.

The study of mendelian forms is decisive in the physiopathological comprehension of AD and related diseases, since the alteration of those genes involved is sufficient to cause the disease. In AD, identification of these genetic causes allows the formulation of the amyloid hypothesis, which is the basis of current therapeutic developments concerning the Ab peptide. Currently three genes (APP, PSEN1, PSEN2) are identified in early onset mendelian forms and their mutations are involved in 80% of the 139 French families, studied since 1993 within the framework of U614 and the National Reference Centre for Alzheimer Disease in young subjects (CNR-MAJ).These results are arguments in favor of the GMAJ project and have two main objectives:

(i) to identify new genes in mendelian AD forms without detectable alteration on known genes.

(ii) to correlate phenotypes and genotypes within families associated with known mutations and extend the description of the phenotypical spectrum.

Population: Families eligible for this study are those with at least 2 individuals with AD criteria (clinical or neuropathological) with onset before 65 years of age. Duration of inclusion is 3 years. This multicentre study groups 23 clinical centres. The inclusion number is 50 new families per year.

Method: Extension and description of families with unknown genetic causes, inclusion of novel families with autosomal dominant AD. The successive steps of the project are the following:

(i) Thorough phenotypical characterization in order to document family history and characterize the probands and affected related subjects according to standardized protocol for clinical, neuropsychological, biological (biomarker determination in plasma and cerebrospinal fluid) and imaging data (MRI, TEMP).

(ii) Identify known genetic causes (PSEN1/2, APP) with novel autosomal dominant families.

(iii) Extend analysis of the pedigrees of families with unknown genetic causes.

(iv) Identify novel genetic causes within these families which are negative for known mutations.

This study uses 3 methods:

* pangenomic search is performed for microalterations (Copy Number Variants or CNV) by Comparative Genomic Hybridization (CGH) with high resolution (10 kb on average).
* potential targets are then validated by the study of large control populations, intrafamilial cosegregation and functional validation.
* the remaining families at the end of this stage will be characterized by means of high throughput sequencing of all exonic areas.

  (v) Follow up study of patients and siblings with 2 goals:
* evaluation of the disease course and consequences (individual, familial and social);
* occurrence of novel AD cases within the family.

(vi) Neuropathological description with potential novel description of atypical AD cases.

Results and consequences: Identification of novel genetic causes of AD are of importance in completing the mechanisms of the amyloidergic hypothesis. This project is useful to promote the guidelines on the genetic diagnosis of AD in France.

ELIGIBILITY:
Inclusion Criteria:

* > in one family 2 cases of Alzheimer disease with age of onset under 65

Exclusion Criteria:

* other cases of young onset dementia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cases of familial Alzheimer disease with age of onset under 65
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2009-11-15 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Didier HANNEQUIN, Pr, Principal Investigator — University Hospital, Rouen
Locations (1):
- CMRR Rouen University Hospital, Rouen, France